CLINICAL TRIAL: NCT01571076
Title: Prospective and Randomized Study of the Use of Comparative Genomic Hybridization (CGH) Arrays to Study Embryo Aneuploidies in Female Advanced Age and Male Factor In Vitro Fertilization (IVF) Patients.
Brief Title: Preimplantation Genetic Screening (PGS) in Advanced Female Age and Male Severe Factor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Carlos Simon, Director of Clinical Research IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1112-C-091-CR
Record Dates: First submitted 2012-03-29; First posted 2012-04-04 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2019-04

CONDITIONS: Embryo Aneuploidies; Implantation Rates; Infertility
Keywords: PGS; CGH; Aneuploidy; Advanced maternal age; Male factor
MeSH Terms: conditions — Infertility; Aneuploidy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group B - Severe Male Factor (Experimental): PGS of day three biopsies and consequent embryo transfer on on Day 5 (blastocyst)
  Interventions: Other: Prolonged culture
- Group B - Advanced Age (Experimental): PGS of day three biopsies and consequent embryo transfer on on Day 5 (blastocyst)
  Interventions: Other: Prolonged culture
- Group A - Advanced Age (Active Comparator): Prolonged culture, no PGS, for Day 5 (blastocyst) embryo transfer for the Advanced Age group
  Interventions: Genetic: PGS
- Group A - Severe Male Factor (Active Comparator): Prolonged culture, no PGS, for Day 5 (blastocyst) embryo transfer for the Severe Male Factor group.
  Interventions: Genetic: PGS

INTERVENTIONS:
Genetic: PGS — Preimplantation Genetic Screening of the embryos and posterior transfer of ongoing Day 5 blastocysts.
  Arms: Group A - Severe Male Factor
Genetic: PGS — Preimplantation Genetic Screening of the embryos and posterior transfer of ongoing Day 5 blastocysts.
  Arms: Group A - Advanced Age
Other: Prolonged culture — The embryos will be in prolonged culture and on going embryos transferred on Day 5 .
  Arms: Group B - Advanced Age
Other: Prolonged culture — Prolonged culture of the embryos and posterior transfer of ongoing Day 5 blastocysts.
  Arms: Group B - Severe Male Factor

SUMMARY:
Preimplantation Genetic Screening (PGS) is used for the selection of chromosomally normal embryos before the transfer in IVF treatments in many cases. There is great debate in the scientific community as to whether this is an efficient practice in patients of different prognosis.

This prospective and randomized study seeks to study the results of chromosomal diagnosis using the new Comparative Genomic hybridization (CGH) arrays technique by practicing Preimplantation Genetic Screening (PGS) in day three biopsy on one arm of the study and not on the other arm in order to compare the results. The investigators will study the ongoing pregnancy rate of each oocyte retrieval and the ongoing implantation rate with Day 5 embryos (blastocysts) in IVF/ intracytoplasmic sperm injection (ICSI) treatments of embryos from two different groups of patients: Advanced Age Female Patients (38 - 41 years of age) and Male severe factor (≥2 million spermatozoids/ml.).

DETAILED DESCRIPTION:
The randomized controlled trial results of advanced maternal age was completed and published (Rubio et al., Fertility&Sterility 2017).

The randomized controlled trial results of the male factor indication was terminated with anticipation due to the change of the technology that prevented recruitment of patients using the old technology (that one used in the study).

ELIGIBILITY:
Inclusion Criteria: ADVANCED AGE and SEVERE MALE FACTOR:

* Women's Age: 38- 41 years old (both included)
* Men's Age: 18-60 years old (both included)
* Ovulation triggered with human chorionic gonadotrophin (hCG) (Ovitrelle, Merck-Serono, Madrid)
* Number of Oocytes metaphase II (MII): ≥ 5 (fresh, not vitrified)
* Quality of semen: ≥ 5 millions spermatozoids/ml

Exclusion Criteria: ADVANCED AGE and SEVERE MALE FACTOR:

* Number of Oocytes metaphase II (MII): <5 oocytes
* Number of Oocytes obtained: >20
* Estradiol on the day of human chorionic gonadotrophin (hCG) >3000 pgr/ml administration.
* Progesterone on the day of hCG >1,5 pmol/l administration
* ≥ 2 previous miscarriages:biochemical,clinical,ectopic or a combination)
* Any un corrected alteration in a previous study.
* Other indications of (Preimplantation Genetic Diagnosis.Screening) PGD-S, such as monogenic illnesses, translocations, repeated implantation failure, repeated miscarriages, etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Ongoing Implantation and Pregnancy Rate | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simon, MDPhD, Principal Investigator — Director; Carmen Rubio, PhD, Study Chair — Igenomix
Locations (1):
- SPAIN: IVI Valencia, IVI Barcelona, IVI Madrid, Valencia, Spain

REFERENCES:
- [Derived] Dahdouh EM, Balayla J, Garcia-Velasco JA. Impact of blastocyst biopsy and comprehensive chromosome screening technology on preimplantation genetic screening: a systematic review of randomized controlled trials. Reprod Biomed Online. 2015 Mar;30(3):281-9. doi: 10.1016/j.rbmo.2014.11.015. Epub 2014 Dec 11. PMID 25599824